CLINICAL TRIAL: NCT02435914
Title: Safety, Efficacy, Tolerability and Pharmacokinetics of AGN-223575 Ophthalmic Suspension in Patients With Dry Eye Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 223575-002
Record Dates: First submitted 2015-05-01; First posted 2015-05-06 (Estimated); Results first posted 2019-04-05 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-03

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- AGN-223575 Dose A (Experimental): 1 drop of AGN-223575 Dose A ophthalmic solution administered in each eye twice daily for 14 day followed by either 1 drop of AGN-223575 Dose A ophthalmic solution or 1 drop of vehicle to AGN-223575 in each eye once daily for 7 days.
  Interventions: Drug: AGN-223575 ophthalmic solution; Drug: AGN-223575 vehicle ophthalmic solution
- AGN-223575 Dose B (Experimental): 1 drop of AGN-223575 Dose B ophthalmic solution administered in each eye twice daily for 14 day followed by either 1 drop of AGN-223575 Dose B ophthalmic solution or 1 drop of vehicle to AGN-223575 in each eye once daily for 7 days.
  Interventions: Drug: AGN-223575 ophthalmic solution; Drug: AGN-223575 vehicle ophthalmic solution
- AGN-223575 Dose C (Experimental): 1 drop of AGN-223575 Dose C ophthalmic solution administered in each eye twice daily for 14 day followed by either 1 drop of AGN-223575 Dose C ophthalmic solution or 1 drop of vehicle to AGN-223575 in each eye once daily for 7 days.
  Interventions: Drug: AGN-223575 ophthalmic solution; Drug: AGN-223575 vehicle ophthalmic solution
- AGN-223575 Vehicle (Placebo Comparator): 1 drop of Vehicle to AGN-223575 ophthalmic solution administered in each eye twice daily for 14 day followed by 1 drop of vehicle to AGN-223575 ophthalmic solution in each eye once daily for 7 days.
  Interventions: Drug: AGN-223575 vehicle ophthalmic solution

INTERVENTIONS:
Drug: AGN-223575 ophthalmic solution — AGN-223575 ophthalmic solution once or twice daily
  Arms: AGN-223575 Dose A; AGN-223575 Dose B; AGN-223575 Dose C
Drug: AGN-223575 vehicle ophthalmic solution — Vehicle to AGN22375 ophthalmic solution once or twice daily.

SUMMARY:
This study will evaluate the safety, efficacy, tolerability, and systemic pharmacokinetics of 3 different doses of topical ophthalmic AGN-223575 suspension compared to AGN-223575 vehicle in patients with dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Signs and symptoms of dry eye disease
* Has used RESTASIS and/or artificial tears in both eyes twice a day for at least 60 days.

Exclusion Criteria:

* History of glaucoma, or ocular hypertension
* Diagnosis of ocular infection
* Use of contact lenses in the past 14 days or expected use during the study
* Use of any topical ophthalmic medications in the past 30 days
* Use of corticosteroids in the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2015-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (28):
- United States (28):
  - Arizona Center for Clinical Trials, Phoenix, Arizona
  - Specialty Eye Ctr. Med. Group, Glendale, California
  - The Eye Research Foundation, Newport Beach, California
  - WCCT Global, Santa Ana, California
  - Eye Associates of Colorado Springs, Colorado Springs, Colorado
  - West Coast Eye Institute, Lecanto, Florida
  - Eye Care Centers Management, Inc., Morrow, Georgia
  - Coastal Research Assoc. LLC, Roswell, Georgia
  - Chicago Cornea Consultants, Hoffman Estates, Illinois
  - Durrie Vision, Overland Park, Kansas
  - Kentucky Center for Vision, Lexington, Kentucky
  - Tufts Medical Center/ Tufts University School of Medicine, Boston, Massachusetts
  - Moyes Eye Center, Kansas City, Missouri
  - Ophthalmology Associates, St Louis, Missouri
  - Comprehensive Eye Care Ltd., Washington, Missouri
  - Raymond Fong MD, PC, New York, New York
  - South Shore Eye Care LLP, Wantagh, New York
  - SE Clinical Research Associates, LLC/ Charolette Eye Ear Nose, Charlotte, North Carolina
  - Cornerstone Eye Care, High Point, North Carolina
  - Eye Care Associates of Greater Cincinnati, Cincinnati, Ohio
  - Mark A. Terry, MD PC/ Devers Eye Institute, Portland, Oregon
  - Bluestein Custom Vision, Charleston, South Carolina
  - Carolinas Centers for Sight, PC, Florence, South Carolina
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Keystone Clinical Research, Austin, Texas
  - Houston Eye Associates, Houston, Texas
  - Whitsett Vision Group, Houston, Texas
  - Medical Center Opth. Assoc., San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AGN-223575 Dose A | AGN-223575 Dose B | AGN-223575 Dose C | AGN-223575 Vehicle
Started | 58 | 59 | 60 | 59
Completed | 57 | 58 | 59 | 59
Not Completed | 1 | 1 | 1 | 0
Not completed — Ocular Adverse Event | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Other Miscellaneous Reason | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AGN-223575 Dose A | AGN-223575 Dose B | AGN-223575 Dose C | AGN-223575 Vehicle | Total
Number analyzed (Participants) | 58 | 59 | 60 | 59 | 236
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (16.37) | 59.2 (14.74) | 56.6 (16.10) | 54.1 (17.87) | 56.0 (16.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 47 | 39 | 46 | 168
  Male | 22 | 12 | 21 | 13 | 68

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Conjunctival Redness Score in the Study Eye Using a 5-Point Scale
Description: Nasal and temporal bulbar conjunctival hyperemia were graded separately in each eye by the investigator under slit-lamp magnification by assigning a score of 0 to 4 for each quadrant based on comparison to the Allergan Dry Eye Redness Scale with photographic reference where: 0=Normal, vessels of bulbar conjunctiva are easily observed; 1=Trace redness; 2=Mild redness; 3=Moderate redness; 4=Severe redness, and each score is associated with a reference photo. For each eye, the study quadrant was determined by the greater (more severe) of the baseline redness scores for nasal and temporal bulbar conjunctival hyperemia as assessed using the Allergan Dry Eye Redness Scale. If the temporal score was greater than the nasal score, then the temporal quadrant was the study quadrant for the eye and was used to assess primary efficacy; otherwise the nasal quadrant was the study quadrant. A negative change from baseline (less redness) indicates improvement.
Time Frame: Baseline, Day 14
Population: Modified Intent-to-treat (mITT) population, consisted of all randomized and treated patients who had a baseline and at least 1 post-baseline assessment of nasal or temporal redness using the Allergan Dry Eye Redness Scale. "n" in the category is the number of participants with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AGN-223575 Dose A | AGN-223575 Dose B | AGN-223575 Dose C | AGN-223575 Vehicle
Number analyzed (Participants) | 58 | 59 | 60 | 57
score on a scale
  Baseline | 1.9 (0.68) | 2.2 (0.69) | 2.0 (0.70) | 2.1 (0.72)
  Change from Baseline at Day 14: number analyzed (Participants) | 56 | 58 | 60 | 57
  Change from Baseline at Day 14 | -0.7 (0.80) | -0.9 (0.76) | -0.8 (0.76) | -0.6 (0.84)

2. Secondary Outcome: Change From Baseline in Ocular Surface Disease Index (OSDI) Total Score Using a 5-Point Scale
Description: OSDI questionnaire consists of 12 questions regarding ocular symptoms, environmental triggers, and vision-related functioning in patients with dry eye disease. The participants rate each question on a 5-point scale where: 0=none of the time to 4=all of the time. The scores are totaled over the 12 questions and normalized/converted to a total score of 0=no disability to 100=complete disability. Higher OSDI scores are associated with greater severity. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Day 14
Population: mITT population, consisted of all randomized and treated participants who had a baseline and at least 1 post-baseline assessment of nasal or temporal redness using the Allergan Dry Eye Redness Scale. "n" in the category is the number of participants with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AGN-223575 Dose A | AGN-223575 Dose B | AGN-223575 Dose C | AGN-223575 Vehicle
Number analyzed (Participants) | 58 | 59 | 60 | 59
score on a scale
  Baseline | 49.65 (16.510) | 51.00 (18.908) | 48.95 (16.472) | 52.63 (19.204)
  Change from Baseline at Day 14: number analyzed (Participants) | 56 | 58 | 60 | 59
  Change from Baseline at Day 14 | -14.64 (16.647) | -15.92 (16.329) | -15.27 (17.305) | -14.76 (17.297)

3. Secondary Outcome: Change From Baseline in Corneal Staining Score of the Study Eye Using a 6-Point Scale
Description: The cornea is the transparent front part of the eye which covers the iris and pupil. Staining of the cornea following ocular administration of fluorescein dye was graded using a 6-point scale where: 0=no staining to 5=diffuse staining. The higher the grade score, the worse the dry eye severity. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AGN-223575 Dose A | AGN-223575 Dose B | AGN-223575 Dose C | AGN-223575 Vehicle
Number analyzed (Participants) | 58 | 59 | 60 | 59
score on a scale
  Baseline | 1.7 (0.76) | 1.9 (0.85) | 1.8 (0.88) | 1.8 (0.75)
  Change from Baseline at Day 14: number analyzed (Participants) | 56 | 58 | 60 | 57
  Change from Baseline at Day 14 | -0.6 (0.82) | -0.6 (0.80) | -0.6 (0.97) | -0.5 (0.89)

4. Secondary Outcome: Percentage of Participants With Complete Redness Response (Yes/No) in the Study Eye
Description: A participant was considered a redness responder if the study quadrant redness score based on the Allergan Dry Eye Redness Scale in the study eye was 0=Normal (no redness).
Time Frame: Day 14
Population: Participants from the mITT population, all randomized and treated participants who had a baseline and at least 1 post-baseline assessment of nasal or temporal redness using the Allergan Dry Eye Redness Scale. with data available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | AGN-223575 Dose A | AGN-223575 Dose B | AGN-223575 Dose C | AGN-223575 Vehicle
Number analyzed (Participants) | 56 | 58 | 60 | 57
percentage of participants
  Yes | 10.7 | 12.1 | 15.0 | 10.5
  No | 89.3 | 87.9 | 85.0 | 89.5

ADVERSE EVENTS:
Arm/Group | AGN-223575 Dose A | AGN-223575 Dose B | AGN-223575 Dose C | AGN-223575 Vehicle
Serious Adverse Events (participants affected / at risk) | 1/58 | 1/59 | 1/60 | 0/59
Other Adverse Events (participants affected / at risk) | 3/58 | 4/59 | 4/60 | 6/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AGN-223575 Dose A (N=58) | AGN-223575 Dose B (N=59) | AGN-223575 Dose C (N=60) | AGN-223575 Vehicle (N=59)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AGN-223575 Dose A (N=58) | AGN-223575 Dose B (N=59) | AGN-223575 Dose C (N=60) | AGN-223575 Vehicle (N=59)
Instillation site pain (General disorders) | 3 | 4 | 4 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.